CLINICAL TRIAL: NCT02042261
Title: The Role of Therapeutic Drug Monitoring in Tuberculosis - a Pilot Study
Status: Completed | Type: Observational
Sponsor: Thomas Schon (Other Government)
Collaborators: University Hospital, Linkoeping (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Thomas Schon, MD PhD, Linkoeping University
Organization: Linkoeping University (Other Government)
Other Study IDs: TB-TDM
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Active Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Drug resistant TB is increasing and in order to enchance the efficacy of the current drugs, individualized therapy using plasma drug concentrations and minimal inhibitory concentration (MIC) determination may be of importance. This concept is defined as therapeutic drug monitoring (TDM).

In this pilot study our hypothesis is that the ratio between MIC and drug concentration data is correlated to the bacterial load measured as time to positive liquid culture (TTP).

In two sites in Sweden (Linköping and Karolinska Hospital Solna, Stockholm), 25 patients with pulmonary tuberculosis will be recruited. MIC-determination of Mycobacterium tuberculosis will be performed in BACTEC 960 MGIT and drug concentration will be determined at 2, 4 and 12 weeks after treatment initiation using LC-MS/MS methodology. Sputum cultures will be obtained at 0, 2 days, 7 days, 2 weeks, 4 weeks and 8 weeks and TTP will be measured in duplicate samples. Clinical follow up according to WHO criteria will be performed 1 year after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

Age>18 years, culture verified tuberculosis

Exclusion Criteria:

Other infectious diseases other than HIV or tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with culture verified tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2012-01; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Rifampicin concentration in relationship to MIC over 10 | 2 weeks

SECONDARY OUTCOMES:
Cure rate on Clinical follow up (according to WHO criteria) in relation to rifampicin concentration at week 2 | 1 year
Sputum Culture conversion in relation to rifampicin, isoniazid and pyrazinamid concentration week 2 | 2 and 8 weeks
TB-score in relation to rifampicin, isoniazid and pyrazinamid concentration week 2 | 8 weeks
Time to positive Culture (TTP) in relation to isoniazid, ethambutol and pyrazinamid serum concentration and minimal inhibitory concentration (MIC) | 2 and 8 weeks
Time to positive Culture (TTP) in relation to rifampicin serum concentration and minimal inhibitory concentration (MIC) | 2weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Niward, MD, Principal Investigator — Linkoeping University
Locations (2):
- Sweden (2):
  - Dept of Infectious Diseases, Linköping, Linköping
  - Dept of Infectious Diseases, TB-unit, Karolinska Hospital, Stockholm, Stockholm County

REFERENCES:
- [Derived] Niward K, Davies Forsman L, Bruchfeld J, Chryssanthou E, Carlstrom O, Alomari T, Carlsson B, Pohanka A, Mansjo M, Jonsson Nordvall M, Johansson AG, Eliasson E, Werngren J, Paues J, Simonsson USH, Schon T. Distribution of plasma concentrations of first-line anti-TB drugs and individual MICs: a prospective cohort study in a low endemic setting. J Antimicrob Chemother. 2018 Oct 1;73(10):2838-2845. doi: 10.1093/jac/dky268. PMID 30124844